CLINICAL TRIAL: NCT00493610
Title: Use of Mucomyst (NAC) to Ameliorate Oxidant Stress as Measured by Surrogate Serum in Patients With Hepatitis C
Brief Title: Mucomyst for Hepatitis C
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaborator no longer interested, short of funds
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: West Virginia University (Other)
Responsible Party: Saklayen, Mohammad - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0031
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis C
Keywords: Oxidant stress; N-acetylcysteine; Hepatitis C; Liver disease; Mucomyst; Isoprostane
MeSH Terms: conditions — Hepatitis C; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: N-acetylcysteine(Mucomyst)

INTERVENTIONS:
Drug: N-acetylcysteine(Mucomyst)

SUMMARY:
The study will examine the effects of treatment with N-acetylcysteine ( Mucomyst ) 1 gm twice a day for 30 dyas in 15 patients with hepatitis C. The primary outcome of interest wil be the changes in oxidant stress as measured by different oxidant stress markers level in sera. Secondary outcomes of interest will be changes in viral load of hep C and changes in liver function

DETAILED DESCRIPTION:
The Effects of N-Acetylcysteine on Oxidative Stress in Chronic Hepatitis C

Objective:

There is evidence that suggests oxidative stress plays a role in the pathologic mechanism of disease progression in chronic hepatitis C virus infection (HCV). This study will test the hypothesis that N-acetylcysteine given over one month will decrease oxidative stress and thus slow disease progression.

Background:

Chronic hepatitis C is the most common blood borne infection in the United States. An average of 230,000 new infections occurred each year during the 1980s, although since 1989 the annual number of new infections has declined by greater than 80% to 36,000 by 1996.1,2,3 A CDC survey in 2003 showed that annual new cases had declined to 30,000.4 The Third National Health and Nutrition Examination Survey (NHANES III), conducted during 1988-1994, indicated that an estimated 3.9 million (1.8%) Americans have been infected with HCV. In the general population, the highest prevalence rates of HCV infection are found among persons aged 30-49 years and among males. Unlike the racial/ethnic pattern of acute disease, African Americans have a substantially higher prevalence of HCV infection than do whites.5 Population-based studies indicate that 40% of chronic liver disease is HCV-related, resulting in estimated deaths of 8,000-10,000 each year. According to the CDC, estimated medical and work-loss costs of HCV-related acute and chronic liver disease are greater than $600 million annually, and HCV-associated end-stage liver disease is the most frequent indication for liver transplantation among adults.1

After an acute infection, chronic HCV infection develops in most persons (75%-85%). 6 The course of chronic HCV is insidious, progressing at a slow rate without symptoms or physical signs in the majority of patients during the first two or more decades. Cirrhosis develops in 10%-20% of persons with chronic HCV over a period of 20-30 years, and hepatocellular cancer in 1%-5%.7

HCV replicates in the hepatocytes, but it is not directly hepatotoxic. Lymphocytes recognize infected cells and initiate an immune response. Damage to the liver parenchyma is mediated by inflammatory cytokines, although the mechanism of disease progression is not clearly understood. Jain et al. and Pratico et al. have shown that oxidative stress may be a factor in progression to fibrosis and cirrhosis.8,9 It is believed that oxidative stress occurs via various mechanisms including the reduction of NAD to NADH that causes a redox change and inhibition of xanthine dehydrogenase activity resulting in a shift of purine oxidation to xanthine oxidase, thereby promoting the generation of oxygen-free radical species. A depletion in glutathione (GSH) has also been found in chronic liver disease which impairs defense against oxidative stress.10 Several other studies have attempted to evaluate for oxidative stress associated with HCV, but until recently accurate markers for evaluation of oxidative stress had not been determined. Studies attempting to treat chronic HCV with interferon and antioxidant combination have been inconclusive due inability to appropriately measure oxidative stress.11, 12

Guha et al. discuss that for a long time, assessment of lipid peroxidation in vivo was restricted to tissue measurements of alkanes, malondialdehyde, or hydroxynonenal levels, all of which have serious limitation in accurately assessing oxidative stress. Roberts and coworkers discovered a series of novel prostaglandins, now termed F2-isoprostanes, which are now considered the gold standard for assessment of oxidative injury in vivo. These prostaglandins are formed initially in situ by oxidation of arachidonic acid containing phospholipids, and then released by the action of phospholipase. These can be measured in plasma or urine samples by using gas chromatography mass spectrometry or ELISA.13-16 Recently, Dr. Vallyathan's group in West Virginia demonstrated that total antioxidant status, glutathione peroxidase, and isoprostane levels were increased in shipyard welders consistent with oxidative stress secondary to their occupational exposures.17

N-acetylcysteine (NAC) is a precursor of reduced GSH. It is an acetylated form of amino acid L-cysteine, and is an excellent source of sulfhydryl groups. It is converted in the body into metabolites capable of stimulating GSH synthesis, promoting detoxification, and acting directly as free radical scavengers. It has been used clinically for more than 30 years primarily as a monolithic. It is now commonly used for pre-treatment to prevent renal injury secondary to intravenous dye in patients with renal insufficiency. It is also a mainstay of treatment in cases of acetaminophen overdose since the 1980s. In this time period, NAC has been shown to be safe without any significant toxicity or side-effects.18 Other studies have shown that NAC can prevent apoptosis and promote cell survival. It reduces endothelial dysfunction, inflammation, fibrosis, cartilage erosion, and transplant prolongation.19 It has also been useful in improving ischemia-reperfusion related liver injury, cocaine and methanol related liver injury.20-23

Considering the above information, it would be worthwhile to evaluate the baseline oxidative stress in patients with hepatitis C and note changes, if any after NAC treatment for 6 months. There have been no prospective studies thus far that have evaluated baseline oxidative stress in Hep C patients on and off interferon treatments with evaluation of F2-isoprostanes and followed up on lab markers after treatment with NAC.

Research design:

Ten patients with HCV proven by PCR, not on treatment, will be recruited from the VA GI clinic patient population. Background data will be gathered from the charts and by a questionnaire. Blood for baseline liver function tests including serum ferritin, serum isoprostane, serum aconitase, plasma glutathione (GSH), glutathione peroxidase (GPx) and total antioxidant status (TAS), will be obtained in all patients. These tests will be repeated in each patient after 15 days and 1 month of NAC at 1000 mg by mouth twice a day. Tests will again be repeated 30 days after stopping the study medication. Hep c mRNA will be measured at baseline and at 30 days. The research protocol will be explained to the patient and informed consent will be obtained prior to enrollment. For the volunteers travel expenses and time, $25 will be given at the beginning and end of the study for participation.

Inclusion criteria will be as follows: Volunteers will be divided into 2 groups: healthy patients and HCV patients not on interferon. Exclusion criteria will be as follows: significantly decompensated liver cirrhosis of Child's Class C, patients with evidence of liver mass or hepatocellular cancer. Patients who are pregnant or on antioxidant such at Vitamin E or Vitamin C will also be excluded. Also patients with known allergy to N-acetylcysteine will be excluded

Sample Size calculation:

Since each patient will be his own control ( reducing the potential confounding of age,

smoking, medicine, life style etc )assuming variance of 5% in the assay system of the biomarkers, 15 patients will give 90% power to see 10% or more difference in aggregate level of the oxidant biomarkers.

Statistical Analyses:

Baseline demographic (age, sex) and clinical data (symptoms, Child's Classification) will be collected for each patient. This data will be compared between the three groups using Student's t-test for continuous variables and either Chi-square or Fisher's exact tests for non-parametric variables. The measured laboratory values in the three groups, for the baseline and post N-acetylcysteine, will be compared by using the paired t-test.

ELIGIBILITY:
Inclusion Criteria:

- Patient with known hepatitis C

Exclusion Criteria:

* Patient on another therapy for Hep C
* Patient on dialysis
* Patient who are allergic to Mucomyst

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Measurable oxidant stress | 30 days

SECONDARY OUTCOMES:
Reduction in viral load of Hep C and changes in Liver Function tests | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad G. Saklayen, MD, Principal Investigator — VA Medical Center, Dayton
Locations (1):
- VA Medical Center, Dayton, Dayton, Ohio, United States